CLINICAL TRIAL: NCT07393321
Title: A Randomized, Double-blind, Placebo-controlled Phase III Trial to Evaluate the Efficacy and Safety of NTQ1062 in Combination With Fulvestrant Versus Placebo Plus Fulvestrant in Patients With Locally Advanced (Unresectable) or Metastatic HR+/HER2- Breast Cancer Who Relapsed or Progressed During or After Endocrine Therapy.
Brief Title: A Phase III Clinical Trial of NTQ1062 in Combination With Fulvestrant for the Treatment of Advanced or Metastatic HR+/HER2- Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTQ1062-301
Record Dates: First submitted 2026-01-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: HR Positive/HER2 Negative Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo+ fulvestrant (Placebo Comparator): Placebo: 200 mg orally twice daily, for 21 consecutive days, followed by 7 days off (21/7 dosing schedule), during a 28-day cycle. Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 and Day 15 of cycle 1, and then on Day 1of each cycle thereafter.
  Interventions: Drug: Placebo + fulvestrant
- NTQ1062+fulvestrant (Experimental): NTQ1062: 200 mg orally twice daily for 21 consecutive days, followed by 7 days off (21/7 dosing schedule), during a 28-day cycle. Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 and Day15 of cycle 1, and then on Day 1 of each cycle thereafter.
  Interventions: Drug: NTQ1062+Fulvestrant

INTERVENTIONS:
Drug: Placebo + fulvestrant — Placebo: 200 mg orally twice daily, for 21 consecutive days, followed by 7 days off (21/7 dosing schedule), during a 28-day cycle.
  Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 and Day 15 of cycle 1, and then on Day 1of each cycle thereafter.
  Arms: placebo+ fulvestrant
Drug: NTQ1062+Fulvestrant — NTQ1062: 200 mg orally twice daily, for 21 consecutive days, followed by 7 days off (21/7 dosing schedule), during a 28-day cycle.
  Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 and Day 15 of cycle 1, and then on Day 1of each cycle thereafter.
  Arms: NTQ1062+fulvestrant

SUMMARY:
NTQ1062-301 is a randomized, double-blind, placebo-controlled Phase III clinical trial to evaluate the efficacy and safety of the small-molecule AKT inhibitor NTQ1062 combined with fulvestrant versus placebo combined with fulvestrant in patients with HR positive, HER2 negative, locally advanced (unresectable) or metastatic breast cancer that has recurred or progressed during or after endocrine therapy and harbors PIK3CA/AKT1/PTEN alterations.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adult female or male subjects who sign the informed consent form and are at least 18 years of age at the time of signing; (2) pre- and/or post-menopausal women are eligible for inclusion. Premenopausal women must receive ovarian function suppression treatment during the study, such as gonadotropin-releasing hormone agonists (GnRHa). Menopause is defined as: prior bilateral oophorectomy; age ≥ 60 years; age < 60 years, with amenorrhea for ≥ 12 months without prior chemotherapy, tamoxifen, toremifene, or ovarian suppression therapy, and follicle-stimulating hormone (FSH) and estradiol levels within the postmenopausal reference range; (3) Histologically confirmed HR positive, HER-2-negative recurrent locally advanced or metastatic breast cancer, as determined by testing of a recent tumor sample; (4) Prior treatment with at least one endocrine therapy regimen (monotherapy or combination therapy, including aromatase inhibitors and selective ER modulators); (5) Subjects must have at least one measurable disease lesion assessable by CT or MRI, or at least one osteolytic or mixed (osteolytic + sclerotic) bone lesion at baseline; (6) Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; (7) No contraindications to fulvestrant, and meets the eligibility requirements for fulvestrant treatment, as assessed by the investigator; (8) Expected survival time of more than 6 months, as assessed by the investigator; (9) Good bone marrow reserve and organ function; (10) Premenopausal women must have a negative pregnancy test before administration and agree to use effective contraception during the trial and for at least 6 months after the last dose.

Exclusion Criteria:

1. unsuitable for endocrine anti-tumor therapy by the investigators, such as symptomatic visceral crises or inflammatory breast cancer that may be life-threatening in the short term;
2. unable to take oral medication, or with severe gastrointestinal disorders that may affect drug absorption, such as intractable nausea and vomiting, chronic diarrhea (diarrhea lasting >4 weeks), or intestinal obstruction;
3. clinically significant glucose metabolism abnormalities, defined as: diagnosed with type 1 diabetes; type 2 diabetes requiring insulin treatment; glycated hemoglobin (HbA1c) ≥8%; fasting blood glucose >9.3 mmol/L in patients with history of type 2 diabetes, or fasting blood glucose >7.0 mmol/L in patients without history of diabetes;
4. prior use of fulvestrant or other selective estrogen receptor degraders (SERDs) or any PI3K/mTOR/Akt inhibitors;
5. other malignancies besides breast cancer within 5 years prior to screening (excluding basal or squamous cell skin cancer, papillary thyroid carcinoma, bladder carcinoma in situ, or cervical carcinoma in situ, or other tumors that have been radically treated and have shown no clinical recurrence for at least 5 years);
6. have undergone major surgery within 28 days prior to the first dose;
7. have participated in other interventional clinical studies of unmarketed products within 28 days prior to the first dose;
8. severe infections requiring systemic intravenous antibiotics within 28 days prior to the first dose;
9. have received >30% bone marrow radiotherapy or extensive radiotherapy within 28 days prior to the first dose, or palliative local radiotherapy (such as thoracic spine and rib radiotherapy) within 14 days prior to the first dose;
10. have received chemotherapy, endocrine therapy, CDK4/6 inhibitors, traditional Chinese medicine with clear anti-tumor indications, or other small molecule targeted anti-tumor drugs within 14 days prior to the first dose or within 5 half-lives of the drug (whichever is shorter);
11. Received potent CYP3A inhibitors or potent CYP3A inducers within 14 days before the first dose;
12. Previous anti-tumor treatment-related toxicities have not recovered to ≤ grade 1 (assessed according to CTCAE 5.0 criteria, excluding indicators required by the inclusion criteria and toxicities judged by the investigator to pose no safety risk, such as alopecia, grade 2 peripheral neuropathy, and hypothyroidism stabilized by hormone replacement therapy);
13. Known active central nervous system (CNS) metastases, including symptomatic brain metastases, leptomeningeal metastases, or spinal cord compression. Patients who are asymptomatic or stable after treatment and do not require steroid treatment are eligible for enrollment, provided that imaging studies during the screening period confirm no progression for at least 4 weeks;
14. History of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease;
15. History of severe cardiovascular or cerebrovascular disease;
16. active hepatitis, defined as positive for hepatitis B surface antigen (HBsAg) and HBV DNA titer above the local laboratory's lower limit of detection; or positive for hepatitis C virus (HCV) antibody and HCV RNA above the local laboratory's lower limit of detection;
17. History of positive human immunodeficiency virus (HIV) test or positive HIV antibody test result;
18. Clinically uncontrollable pleural, abdominal, or pericardial effusion requiring repeated drainage at the time of screening;
19. Allergy to any active or inactive ingredient of NTQ1062, fulvestrant, or LHRH agonists;
20. Presence of pre-existing or concomitant diseases that the investigator believes may interfere with trial compliance;
21. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as assessed by investigators according to RECIST v1.1 | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter.
  Progression-free survival (PFS) as assessed by investigators according to RECIST v1.1, defined as the time from randomization to the date of disease progression or death from any cause.

SECONDARY OUTCOMES:
PFS assessed by BICR according to RECIST v1.1. | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter.
  PFS assessed by BICR according to RECIST v1.1.
Overall survival (OS) defined as the time from randomization to the date of death from any cause. | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter.
Duration of response (DoR), defined as the time from the date of first recorded response to the date of documented disease progression or the date of death in the absence of documented progression. | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter
Disease control rate (DCR), defined as the percentage of subjects achieving CR, PR, or stable disease (SD) per RECIST v1.1 | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter.
Clinical benefit rate (CBR), defined as the percentage of patients achieving CR, PR, or stable disease (without subsequent anticancer therapy) per RECIST v1.1 | From date of inclusion until the date of first documented progression, assessed up to 60 months. Assessed every 8 weeks for the first 12 months and every 12 weeks thereafter.